CLINICAL TRIAL: NCT05857956
Title: A Clinical Trial to Assess the Efficacy of a Plant-based Energy Shot on Focus and ADHD-like Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proper Wild, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20290
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: ADHD; Attention Difficulties; Mood; Anxiety; Caffeine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proper Wild energy shot (Experimental): Participants will take one bottle daily of Proper Wild Energy shot in the morning. Participants will be advised to drink one bottle in the morning, with or without a meal, depending on their preference, as a replacement for their usual first caffeinated beverage of the day.
  Interventions: Other: Proper Wild energy shot

INTERVENTIONS:
Other: Proper Wild energy shot — 100% plant-based energy shot containing natural caffeine, L-Theanine, purified water, pineapple juice concentrate, natural flavors, kiwi juice concentrate, organic lemon juice concentrate, organic strawberry juice concentrate, monk fruit juice concentrate, pink himalayan sea salt.

SUMMARY:
This is a virtual, single-arm clinical trial that will last 28 days. Participants will drink 1 bottle of Proper Wild energy shot daily and complete questionnaires at baseline, day 1, day 14, and day 28.

Attention deficit hyperactivity disorder (ADHD)-like symptoms, such as concentration, focus, and attention, will be evaluated at baseline and at each check-in. Likert scale responses will be examined from baseline to each check-in. Participant responses on product feedback will be presented as % scores.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing symptoms associated with ADHD, including:

Impulsiveness. Disorganization and problems prioritizing Poor time management skills Problems focusing on a task Trouble multitasking Excessive activity or restlessness Poor planning

* Age 18-55
* Self-reported issues with focus and/or productivity
* Generally healthy - don't live with any uncontrolled chronic disease

Exclusion Criteria:

* Currently taking prescription medication for ADHD
* Currently supplementing with L-Theanine.
* Known to respond negatively to caffeine (no effect, makes them sleepy or feel unwell)
* People with a high caffeine tolerance defined as regular consumption of >400mg of caffeine (>4 coffees) per day.
* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with known severe allergic reactions.
* Women who are pregnant, breastfeeding, or attempting to become pregnant
* Unwilling to follow the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Attention-deficit/hyperactivity disorder (ADHD)-like symptoms. [Time Frame: Baseline to Day 28] | 28 days
  Survey-based assessment (0-5) scale of changes in symptoms associated with ADHD. Parameters explored include focus & concentration, productivity, mood, and "brain fog".

SECONDARY OUTCOMES:
Assess the product as a replacement for coffee or caffeinated beverages. [Time Frame: Baseline to Day 28] | 28 days
  Survey-based assessment regarding changes in daily coffee/beverage consumption, stress, anxiety, jitters, energy crash, and gastrointestinal upset. Responses will be statistically analyzed and reported as % of subject responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided